CLINICAL TRIAL: NCT02265731
Title: A Phase 1/2 Study Evaluating the Safety, Pharmacokinetics and Efficacy of Venetoclax in Japanese Subjects With Hematological Malignancies
Brief Title: Study Evaluating Venetoclax in Subjects With Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-834
Record Dates: First submitted 2014-10-15; First posted 2014-10-16 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Non-Hodgkin Lymphoma (NHL); Multiple Myeloma (MM); Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Acute Myeloid Leukemia (AML)
Keywords: relapsed multiple myeloma; refractory multiple myeloma; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Lymphatic Diseases; relapsed chronic lymphocytic leukemia; small lymphocytic lymphoma; relapsed small lymphocytic lymphoma; refractory small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; acute myeloid leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Lymphoproliferative Disorders; Lymphatic Diseases | interventions — venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Phase 1) (Experimental): Step-up doses of venetoclax to the designated cohort dose administered in participants with relapsed or refractory (R/R) Non-Hodgkin lymphoma (NHL) or multiple myeloma (MM)
  Interventions: Drug: venetoclax
- Arm B (Phase 1) (Experimental): Step-up doses of venetoclax to the designated dose administered in participants with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL)
  Interventions: Drug: venetoclax
- Arm C (Phase 1) (Experimental): Step-up doses of venetoclax to the designated dose with the addition of azacitidine administered in participants with acute myeloid leukemia (AML)
  Interventions: Drug: azacitadine; Drug: venetoclax
- Arm D (Phase 2) (Experimental): Step-up doses of venetoclax to the designated dose with the addition of rituximab in participants with R/R CLL
  Interventions: Drug: venetoclax; Drug: rituximab / IDEC-C2B8

INTERVENTIONS:
Drug: azacitadine — 75 mg/m2 by IV infusion or subcutaneous dosing
  Arms: Arm C (Phase 1)
Drug: venetoclax — Step-up doses of venetoclax to the designated cohort dose
Drug: rituximab / IDEC-C2B8 — 375 mg/m2 on Week 6
  Arms: Arm D (Phase 2)
Drug: rituximab / IDEC-C2B8 — 500 mg/m2 Week 10 Day 1 and thereafter
  Arms: Arm D (Phase 2)

SUMMARY:
This study is evaluating the safety, pharmacokinetic profile and efficacy of venetoclax under a once daily dosing schedule in Japanese participants with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically documented diagnosis of NHL (and exhausted options considered standard of care) as defined in the World Health Organization classification scheme and relapsed following or be refractory to standard treatments such as R-CHOP, R-CVP, or fludarabine based regimens. Participants with other lymphoproliferative diseases can be considered in consultation with the AbbVie medical monitor
* Relapsed or refractory multiple myeloma participants must have been previously treated with at least one prior line of therapy and have measurable disease
* Chronic lymphocytic leukemia/small lymphocytic lymphoma participants must have relapsed or be refractory to standard treatments such as fludarabine based regimens or alkylator based regimens
* Untreated AML subjects or Relapsed or refractory AML subjects must have been previously treated with at least one prior line of therapy
* Eastern Cooperative Oncology Group (ECOG) performance score less than or equal to 1; adequate bone marrow independent of growth factor support per local laboratory reference range; and adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening
* Participants with a history of autologous or allogenic stem cell transplantation must have adequate blood counts independent of growth factor support and have recovered from any transplant-related toxicity(s) and be at least 100 days post-autologous transplant (multiple myeloma) or 6 month post-autologous transplant (NHL) prior to first dose of study drug or at least 6 months post-allogenic transplant (multiple myeloma) prior to first dose of study drug and not have active graft-versus-host disease (GVHD), i.e., requiring treatment

Exclusion Criteria:

* NHL participants who have undergone an allogeneic stem cell transplant or were diagnosed with Post-Transplant Lymphoproliferative Disease, Burkitt's lymphoma, Burkitt-like lymphoma, or lymphoblastic lymphoma/leukemia
* Participant tested positive for HIV
* Participant has a cardiovascular disability status of New York Heart Association Class greater or equal to 2
* Participant has a significant history of renal, neurologic, psychiatric, pulmonary, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the Investigator would adversely affect his/her participating in this study.
* Participant received a monoclonal antibody for anti-neoplastic intent within 8 weeks prior to the first dose of study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Number of participants having treatment-emergent adverse events | Approximately 2 years
  Collect all adverse events at each visit
Time to maximum plasma concentration (Tmax) of venetoclax | Approximately 8 days
Maximum plasma concentration (Cmax) of venetoclax | Approximately 8 days
Area under the plasma concentration-time curve from 0 to 24 hours (AUC24) post-dose of venetoclax | Approximately 8 days
Objective Response Rate (Phase 2) | Approximately 48 months
  The proportion of participants with response (e.g., partial, complete response) using IWCLL (International Workshop on Chronic Lymphocytic Leukemia) criteria for CLL participants will be computed for all participants with active disease at baseline (in the opinion of the investigator).

SECONDARY OUTCOMES:
Objective Response Rate (Phase 1) | Approximately 48 months
  The proportion of participants with response (e.g., partial, complete response) using IWG (International Working Group) response criteria for NHL participants, IMWG (International Myeloma Working Group) response criteria for multiple myeloma participants, IWCLL (International Workshop on Chronic Lymphocytic Leukemia) criteria for CLL participants or IWG (International Working Group) criteria for AML participants will be computed for all participants with active disease at baseline (in the opinion of the investigator).
Minimal Residual Disease (MRD) | Approximately 2 years
Duration of Response | Approximately 48 months
  Duration of response is defined as the number of days from the participant's initial response (e.g., partial, complete response per disease-appropriate response criteria) to the day that disease progression is objectively documented.
Time to disease progression | Approximately 48 months
  Time to disease progression is defined as the number of days from the date the subject started the study drug to the date of the subject's progression (all events of progression will be included).
complete response or remission (CR) rate | Approximately 48 months
  CR rate will be defined as the proportion of participants who achieved a complete response or remission (CR) or complete response with incomplete bone marrow recovery or complete remission with incomplete count recovery (CRi) per the 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria.
Partial response or remission (PR) rate | Approximately 48 months
  PR rate will be defined as the proportion of subjects who achieved a nodular PR (nPR) or PR per the 2008 IWCLL criteria.
Progression Free Survival (PFS) | Approximately 48 months
  Duration of progression-free survival (PFS) will be defined as the number of days from the date of first dose to the date of earliest disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (14):
- Japan (14):
  - NHO Nagoya Medical Center /ID# 129222, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 129061, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 129278, Nagoya, Aichi-ken
  - University of Fukui Hospital /ID# 165801, Yoshida-gun, Fukui
  - National Hospital Organization Kyushu Cancer Center /ID# 149741, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 163202, Fukuoka, Fukuoka
  - Kobe City Medical Center General Hospital /ID# 170919, Kobe, Hyōgo
  - Tohoku University Hospital /ID# 129275, Sendai, Miyagi
  - Kindai University Hospital /ID# 169554, Osakasayama-shi, Osaka
  - Osaka University Hospital /ID# 169862, Suita-shi, Osaka
  - National Cancer Center Hospital /ID# 129044, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 129277, Koto-ku, Tokyo
  - Toranomon Hospital /ID# 148229, Minato-ku, Tokyo
  - NTT Medical Center Tokyo /ID# 166281, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Izutsu K, Yamamoto K, Kato K, Ishikawa T, Fukuhara N, Terui Y, Choi I, Humphrey K, Kim SY, Okubo S, Ogawa N, Nishimura Y, Salem AH, Maruyama D. Phase 1/2 study of venetoclax, a BCL-2 inhibitor, in Japanese patients with relapsed or refractory chronic lymphocytic leukemia and small lymphocytic lymphoma. Int J Hematol. 2021 Mar;113(3):370-380. doi: 10.1007/s12185-020-03024-3. Epub 2020 Oct 23. PMID 33094474